CLINICAL TRIAL: NCT00549354
Title: Endologix Bifurcated PowerLink System Clinical Study
Brief Title: Abdominal Aortic/Aorto-Iliac Aneurysm Endoluminal Graft Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arizona Heart Institute (Other)
Collaborators: Endologix (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-005
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2007-10

CONDITIONS: Aortic Aneurysm
Keywords: Abdominal Infrarenal Aortic; Aorto-Iliac Aneurysms
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Endoluminal Graft

SUMMARY:
The Bifurcated PowerLink System is intended to provide a permanent alternative conduit for blood flow within a patient's abdominal vascular system, which excludes the aneurysmal sac from blood flow and pressure.

DETAILED DESCRIPTION:
An arterial anuerysm is a permanent, localized dilatation of an artery with an increase in diameter ≥ 50% larger than the normal artery. Although any artery may develop an aneurysm, they are most commonly seen in the abdominal aorta, the thoracic aorta, the popliteal artery and the common iliac artery.

The use of intravascular stents and endoluminal grafts to exclude natural arterial aneurysms or treat occlusive vascular lesions has been evaluated in a number of preclinical studies. Endovascular stent graft implantation obviates the need for abdominal surgery by using the peripheral arteries as a route to the aneurysm, and stents provide a means of graft attachment other than sutures. The goal of endoluminal grafting is the same as that of conventional repair and allows insertion of a resilient conduit between the ends of the aneurysm to exclude it from the circulation and prevent rupture of the aneurysm.

This is a Phase 2 Clinical Study of the Bifurcated PowerLink System (Endoluminal Graft) for the treatment of abdominal infrarenal aorto-iliac aneurysmal disease (AAA). Diagnostic imaging methods such as Spiral CT Scans, angiography, ultrasound and fluoroscopy imaging will be used to choose the sites for placement of the device and to assure precise deployment.

The Delivery Catheter allows endovascular placement of the Device (endoluminal graft) via either retrograde (femoral or iliac arteries) or antegrade (brachial arteries) approaches. The Endoluminal Graft (ELG) is a self-expanding metal alloy stent cage, which is covered on the outside by a thin walled ePTPE graft material. The graft material is fully supported throughout the entire ELG length. The ELG is also available in a bifurcated configuration. The bifurcated delivery catheter is available in various diameters and working lengths. The catheter consists of an introducer sheath with homeostatic vavle and an inner shaft. The inner shaft is an obturator with a tapered tip connected to a rear obturator by means of a hypotube. The main body of the ELG is compressed around the hypotube then loaded into the Delivery Catheter. The contralateral and ipsilateral limbs of the ELG are compressed in their respective limb covers and loaded into the Delivery Catheter. The inner shaft accommodates a standard .035 inch guidewire.

The concurrent surgical control and test patients' participation in the Study will include enrollment, the Investigational Device procedure or surgical repair and follow-up period. Patient data will be collected during: pre-operative, operative and post-operative follow-up at discharge and at 1 month. Long term follow-up for both the concurrent surgical controls and test patients will continue for 6 and 12 months to support a PMA. Extended follow-up may be required until the Investigational Device is approved under a PMA, or up to 5 years follow-up under Post Market Surveillance requirements.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Informed consent understood and signed
* Will comply with post-treatment follow-up requirements
* Candidate for conventional open surgical repair

Anatomic Inclusion Criteria:

* Aneurysm is ≥ 4.0 cm in outer diameter or Saccular aneurysm ≥ 3.0 cm in outer diameter or Aneurysm ≥ twice the normal aortic outer diameter or rapidly growing aneurysm (≥ 5 mm over 6 months)

Exclusion Criteria:

* Life expectancy < 2 years
* Participating in another clincal research study
* Pregnant or lactating women
* Acutely ruptured or leaking aneurysm, or vascular injury due to trauma
* Patient has other medical or psychiatric problems, which in the opinion of the Investigator, precludes them from participating in the Study.
* Contrast medium or anticoagulation drugs are contraindicated
* Coagulopathy or bleeding disorder
* Active systemic or localized groin infection
* Inferior mesenteric artery is indispensable
* Connective tissue disease (e.g. Marfan's Syndrome)
* Creatinine level > 1.7 mg/dl
* Thrombus at implantation sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2000-08; Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Mortality Rate | one year
Major complications: myocardial infarction, coronary intervention, respiratory failure, aneurysm rupture, kidney failure, stroke or death | one year

SECONDARY OUTCOMES:
Delivery and stent graft deployment success | 1 month, 6 month, and 12 months
Apposition to the vessel wall | 1 month, 6 month, and 12 months
Device Integrity | 1 month, 6 month, and 12 months
Stent graft patency, occlusion (non-patency) and migration | 1 month, 6 month, and 12 months
Duration of surgical procedure and hospitalization | 1 month, 6 month, and 12 months
Time spent in the ICU | 1 month, 6 month, and 12 months
Amount of blood loss and number of patients requiring blood transfusion with stored blood | 1 month, 6 month, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Diethrich, M.D., Principal Investigator — Arizona Heart Institute
Locations (1):
- Arizona Heart Institute, Phoenix, Arizona, United States

REFERENCES:
- [Background] Bickerstaff LK, Hollier LH, Van Peenen HJ, Melton LJ 3rd, Pairolero PC, Cherry KJ. Abdominal aortic aneurysms: the changing natural history. J Vasc Surg. 1984 Jan;1(1):6-12. PMID 6481873
- [Background] Castleden WM, Mercer JC. Abdominal aortic aneurysms in Western Australia: descriptive epidemiology and patterns of rupture. Br J Surg. 1985 Feb;72(2):109-12. doi: 10.1002/bjs.1800720213. PMID 3971115
- [Background] Lilienfeld DE, Gunderson PD, Sprafka JM, Vargas C. Epidemiology of aortic aneurysms: I. Mortality trends in the United States, 1951 to 1981. Arteriosclerosis. 1987 Nov-Dec;7(6):637-43. doi: 10.1161/01.atv.7.6.637. PMID 3689207
- [Background] Bickerstaff LK, Pairolero PC, Hollier LH, Melton LJ, Van Peenen HJ, Cherry KJ, Joyce JW, Lie JT. Thoracic aortic aneurysms: a population-based study. Surgery. 1982 Dec;92(6):1103-8. PMID 7147188
- [Background] McFarlane MJ. The epidemiologic necropsy for abdominal aortic aneurysm. JAMA. 1991 Apr 24;265(16):2085-8. PMID 2013928
- [Background] Collin J, Araujo L, Walton J. How fast do very small abdominal aortic aneurysms grow? Eur J Vasc Surg. 1989 Feb;3(1):15-7. doi: 10.1016/s0950-821x(89)80102-1. PMID 2714450
- [Background] Bernstein EF, Chan EL. Abdominal aortic aneurysm in high-risk patients. Outcome of selective management based on size and expansion rate. Ann Surg. 1984 Sep;200(3):255-63. doi: 10.1097/00000658-198409000-00003. PMID 6465980
- [Background] Delin A, Ohlsen H, Swedenborg J. Growth rate of abdominal aortic aneurysms as measured by computed tomography. Br J Surg. 1985 Jul;72(7):530-2. doi: 10.1002/bjs.1800720709. PMID 4016532
- [Background] Cronenwett JL, Murphy TF, Zelenock GB, Whitehouse WM Jr, Lindenauer SM, Graham LM, Quint LE, Silver TM, Stanley JC. Actuarial analysis of variables associated with rupture of small abdominal aortic aneurysms. Surgery. 1985 Sep;98(3):472-83. PMID 3898453
- [Background] Brown PM, Pattenden R, Gutelius JR. The selective management of small abdominal aortic aneurysms: the Kingston study. J Vasc Surg. 1992 Jan;15(1):21-5; discussion 25-7. doi: 10.1067/mva.1992.33840. PMID 1728677
- [Background] Guirguis EM, Barber GG. The natural history of abdominal aortic aneurysms. Am J Surg. 1991 Nov;162(5):481-3. doi: 10.1016/0002-9610(91)90266-g. PMID 1951914
- [Background] Ouriel K, Green RM, Donayre C, Shortell CK, Elliott J, DeWeese JA. An evaluation of new methods of expressing aortic aneurysm size: relationship to rupture. J Vasc Surg. 1992 Jan;15(1):12-8; discussion 19-20. doi: 10.1067/mva.1992.32982. PMID 1728670
- [Background] Limet R, Sakalihassan N, Albert A. Determination of the expansion rate and incidence of rupture of abdominal aortic aneurysms. J Vasc Surg. 1991 Oct;14(4):540-8. doi: 10.1067/mva.1991.30047. PMID 1920652
- [Background] Nevitt MP, Ballard DJ, Hallett JW Jr. Prognosis of abdominal aortic aneurysms. A population-based study. N Engl J Med. 1989 Oct 12;321(15):1009-14. doi: 10.1056/NEJM198910123211504. PMID 2674715
- [Background] Ingoldby CJ, Wujanto R, Mitchell JE. Impact of vascular surgery on community mortality from ruptured aortic aneurysms. Br J Surg. 1986 Jul;73(7):551-3. doi: 10.1002/bjs.1800730711. PMID 3730787
- [Background] Crawford ES, DeNatale RW. Thoracoabdominal aortic aneurysm: observations regarding the natural course of the disease. J Vasc Surg. 1986 Apr;3(4):578-82. doi: 10.1067/mva.1986.avs0030578. PMID 3959256
- [Background] Dotter CT. Transluminally-placed coilspring endarterial tube grafts. Long-term patency in canine popliteal artery. Invest Radiol. 1969 Sep-Oct;4(5):329-32. doi: 10.1097/00004424-196909000-00008. No abstract available. PMID 5346893
- [Background] Cragg A, Lund G, Rysavy J, Castaneda F, Castaneda-Zuniga W, Amplatz K. Nonsurgical placement of arterial endoprostheses: a new technique using nitinol wire. Radiology. 1983 Apr;147(1):261-3. doi: 10.1148/radiology.147.1.6828742.
- [Background] Maass D, Zollikofer CL, Largiader F, Senning A. Radiological follow-up of transluminally inserted vascular endoprostheses: an experimental study using expanding spirals. Radiology. 1984 Sep;152(3):659-63. doi: 10.1148/radiology.152.3.6463245.
- [Background] Balko A, Piasecki GJ, Shah DM, Carney WI, Hopkins RW, Jackson BT. Transfemoral placement of intraluminal polyurethane prosthesis for abdominal aortic aneurysm. J Surg Res. 1986 Apr;40(4):305-9. doi: 10.1016/0022-4804(86)90191-5. PMID 3702388
- [Background] Lawrence DD Jr, Charnsangavej C, Wright KC, Gianturco C, Wallace S. Percutaneous endovascular graft: experimental evaluation. Radiology. 1987 May;163(2):357-60. doi: 10.1148/radiology.163.2.2951767.
- [Background] Palmaz JC, Sibbitt RR, Tio FO, Reuter SR, Peters JE, Garcia F. Expandable intraluminal vascular graft: a feasibility study. Surgery. 1986 Feb;99(2):199-205. PMID 2935960
- [Background] Palmaz JC, Parodi JC, Barone HD, et al. Transluminal bypass of experimental abdominal aortic aneurysm. RSNA 1990; 177(s):202.
- [Background] Yoshioka T, Wright KC, Wallace S, Lawrence DD Jr, Gianturco C. Self-expanding endovascular graft: an experimental study in dogs. AJR Am J Roentgenol. 1988 Oct;151(4):673-6. doi: 10.2214/ajr.151.4.673. PMID 3262266
- [Background] Mirich D, Wright KC, Wallace S, Yoshioka T, Lawrence DD Jr, Charnsangavej C, Gianturco C. Percutaneously placed endovascular grafts for aortic aneurysms: feasibility study. Radiology. 1989 Mar;170(3 Pt 2):1033-7. doi: 10.1148/radiology.170.3.2916054.
- [Background] Chuter TA, Green RM, Ouriel K, Fiore WM, DeWeese JA. Transfemoral endovascular aortic graft placement. J Vasc Surg. 1993 Aug;18(2):185-95; discussion 195-7. doi: 10.1067/mva.1993.42587. PMID 8350427
- [Background] Laborde JC, Parodi JC, Clem MF, Tio FO, Barone HD, Rivera FJ, Encarnacion CE, Palmaz JC. Intraluminal bypass of abdominal aortic aneurysm: feasibility study. Radiology. 1992 Jul;184(1):185-90. doi: 10.1148/radiology.184.1.1535160.
- [Background] Hagen B, Harnoss BM, Trabhardt S, Ladeburg M, Fuhrmann H, Franck C. Self-expandable macroporous nitinol stents for transfemoral exclusion of aortic aneurysms in dogs: preliminary results. Cardiovasc Intervent Radiol. 1993 Nov-Dec;16(6):339-42. doi: 10.1007/BF02603137. PMID 8131163
- [Background] Parodi JC, Palmaz JC, Barone HD. Transfemoral intraluminal graft implantation for abdominal aortic aneurysms. Ann Vasc Surg. 1991 Nov;5(6):491-9. doi: 10.1007/BF02015271. PMID 1837729
- [Background] Parodi JC. Endovascular repair of abdominal aortic aneurysms and other arterial lesions. J Vasc Surg. 1995 Apr;21(4):549-55; discussion 556-7. doi: 10.1016/s0741-5214(95)70186-9. PMID 7707560
- [Background] May J, White G, Waugh R, Yu W, Harris J. Transluminal placement of a prosthetic graft-stent device for treatment of subclavian artery aneurysm. J Vasc Surg. 1993 Dec;18(6):1056-9. PMID 8264035
- [Background] Cragg AH, Dake MD. Percutaneous femoropopliteal graft placement. Radiology. 1993 Jun;187(3):643-8. doi: 10.1148/radiology.187.3.8497609.
- [Background] Dake MD, Miller DC, Semba CP, Mitchell RS, Walker PJ, Liddell RP. Transluminal placement of endovascular stent-grafts for the treatment of descending thoracic aortic aneurysms. N Engl J Med. 1994 Dec 29;331(26):1729-34. doi: 10.1056/NEJM199412293312601. PMID 7984192
- [Background] Piquet P, Bartoli JM, Rolland PH, Mercier C. Tantalum Dacron co-knit stent for endovascular treatment of aorto-iliac aneurysms. Presented at the 17th World Congress of the International Union of Angiology, London, England, April 1995.
- [Background] Parodi J. Presented at III International Endovascular Surgery Symposium, Sydney, Australia, November 1993 and VII International Congress on Endovascular Interventions, Phoenix, Arizona, February 1994.
- [Background] Moore W. Presented the Southern California Chapter of the American College of Surgeons Meeting, Newport Beach, CA. January 1994.
- [Background] Ahn R. Presented at VII International Congress on Endovascular Interventions, Phoenix, Arizona, February 1994.
- [Background] May J, White GH. Presented at III International Endovascular Surgery Symposium, Sydney, Australia, November 1993 and VII International Congress on Endovascular Interventions, Phoenix, Arizona, February 1994.
- [Background] Chuter T. Presented at III International Endovascular Surgery Symposium, Sydney, Australia, November 1993 and VII International Congress on Endovascular Interventions, Phoenix, Arizona, February 1994.
- [Background] Marin ML. Stented grafts for the treatment of aorto-iliac and femoropopliteal occlusive disease. Abstract, VII International Congress on Endovascular Interventions, Phoenix, Arizona, February 1994.
- [Background] Vieth FJ, Mann ML, Panetta TF, Parodi JC, Cinaron J. Stented grafts for the treatment of traumatic arterial lesions and non-aortic aneurysms. Abstract, VII International Congress on Endovascular Interventions, Phoenix, Arizona, February 1994.
- [Background] Semba CP, Dake MD, Mitchell RS, Miller DC. Endovascular grafting for the treatment of thoracic aortic aneurysms: Preliminary experience at Stanford University Medical Center. Abstract, VII International Congress on Endovascular Interventions, Phoenix, Arizona, February 1994.
- [Background] Diethrich EB, Parazoglou CD, Lundquist P, Rodriguez-Lopez J, Lopez-Galarza L, Eckert J, Stone D, Cassess R, Matveevskii A. Early experience with aneurysm exclusion devices and endoluminal bypass prosthesis. Abstract, VII International Congress on Endovascular Interventions, Phoenix, Arizona, February 1994.
- [Background] Ivancev K, Chuter T, Lindblad B, et al. Endovascular treatment of perigraft perfusion following transfemoral aneurysm repair. World J Surg 1996; in press.
- [Background] Chuter T, Hopinson B, Wendt G et al. Transfemoral aortic aneurysm repair with bifurcated endovascular grafts. Presented at the 43rd meeting of the International Society for Cardiovascular surgery, North American Chapter, New Orleans, LA June 1995.
- [Background] Parodi JC. Endoluminal treatment of aortic aneurysms. Presented at the 2nd International Workshop on Interventional Radiology, Czech Radiological Society, Prague, June 1995.
- [Background] Mailhe C. Results of the Stentor Trial. Presented at the 17th World Congress of the International Union of Angiology, London, England, April 1995.
- [Background] Mann ML. Complications of endovascular stented grafts for the treatment of arterial lesions: The agony after ecstasy. Presented at the 43rd meeting of the International Society for Cardiovascular Surgery, North American Chapter, New Orleans, LA, June 1994.
- [Background] Suggested standards for reports dealing with lower extremity ischemia. Prepared by the Ad Hoc Committee on Reporting Standards, Society for Vascular Surgery/North American Chapter, International Society for Cardiovascular Surgery. J Vasc Surg. 1986 Jul;4(1):80-94. PMID 3723692
- [Background] Ancure Summary of Safety and Efficacy, Table 16, page 18 of 24.
- [Background] AneuRx Summary of Safety and Efficacy. Adverse Events, Section 8, Page 7.